CLINICAL TRIAL: NCT05821049
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Evaluate the Efficacy of UP165 on Sleep Quality and Mood State in Healthy Adults
Brief Title: A Study to Evaluate the Efficacy of UP165 on Sleep Quality and Mood State in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: UI/220902/UP/SQMS
Record Dates: First submitted 2023-03-23; First posted 2023-04-20 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Sleep Disturbance
Keywords: Sleep Quality
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: A randomized, double blind, placebo controlled, parallel group
Who Masked: Participant, Care Provider, Investigator
Masking Description: Envelope Blinding Chits
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UPI65 (Low Dose) (Active Comparator): One capsule to be taken 60 ± 10 mins before bed
  Interventions: Other: UPI65 (Low Dose)
- UPI65 (High Dose) (Active Comparator): One capsule to be taken 60 ± 10 mins before bed
  Interventions: Other: UP165 (High Dose)
- Placebo (Placebo Comparator): One capsule to be taken 60 ± 10 mins before bed
  Interventions: Other: Placebo

INTERVENTIONS:
Other: UPI65 (Low Dose) — Red colored Capsules
  Arms: UPI65 (Low Dose)
Other: UP165 (High Dose) — Red colored Capsules
  Arms: UPI65 (High Dose)
Other: Placebo — Red colored Capsules
  Arms: Placebo

SUMMARY:
A randomized, double blind, placebo controlled, parallel group study to evaluate the efficacy of UP165 on sleep quality and mood state in healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥20 and ≤ 60 years' old with moderate physical activity level as per International Physical Activity Questionnaire - Short Form(IPAQ - SF)
* Volunteers with body mass index between 18.5 and 29.9 kg/m2. Fairly bad or very bad subjective sleep quality with a score of 2 or 3 assessed as per PSQI Q9.
* Willing to maintain current dietary pattern, activity level, and stable bodyweight for the duration of the study, and refrain from any drastic lifestyle changes.
* Unable to fall asleep or unable to stay asleep (2 or more waking episodes during sleep at least twice a week but not more than four times)
* Agrees to maintain current sleep schedule throughout the study
* Agrees to stay in the current time zone for the duration of the study
* Subjects ready to give voluntary, written, informed consent to participate in the study.
* Willing to complete all study procedures including study-related questionnaires and comply with study requirements.

Exclusion Criteria:

* Subjects diagnosed with sleep disorders secondary to another health problem.
* Consumption of hypnotic drugs (<3 months before inclusion).
* Subjects with a history of caffeine consumption post 6:00 pm.
* Individuals taking any other sleep supplements and are unwilling to stop taking those supplements for the duration of the study period
* Recent history of physical, emotional, social trauma within last three months.
* Participants who are not medication (which are likely to impact sleep quality or pattern) free for at least 4 weeks apart from contraceptive pills
* Subjects who consume pain-relieving medications more than once per week.
* Individuals who have night terrors regularly
* Individuals who regularly sleepwalk
* Individuals who work at night shifts.
* Individuals who have regular bad dreams
* Use of the following medications during the study period: oral or injectable corticosteroid, sedating antihistamines (e.g. cold, allergy, motion sickness), psychotropic medications or hypnotics, benzodiazepine, narcotics, any illicit drugs
* Gastro-intestinal, hepatic, respiratory, psychiatric, kidney, or cardiovascular disorder (<3 months before inclusion),
* Recent (<3 months before inclusion) change in lifestyle (food, body weight, sport, drug, and/or dietary supplement),
* Students having regular class and assignments
* Subjects addicted to digital media who exhibit at least five of the following symptoms currently:

  i) Preoccupation with the digital media use j) Withdrawal symptoms that occur when digital media use is not possible k) Build-up of a tolerance that requires increasing amounts of digital media use to satisfy cravings l) Unsuccessful attempts to stop or limit digital media use m) Replacement of previously pleasurable activities with digital media use n) Unwillingness to stop digital media use despite its negative consequences o) Being deceptive about digital media use p) Using digital media use as a coping mechanism
* Addiction or history of substance abuse,
* Consumption of more than 3 glasses of alcohol per day,
* Pregnant or lactating woman,
* Lifestyle habits which would modify the wake-sleep rhythm, or which was expected to be modified during the study period (e.g., night work), and finally,
* Known allergy to the IP.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of the Investigational Product (IP) from baseline on | throughout the study period (approximately 28 days)
  Sleep statistics (sleep quality thoughout the study) by using the watch known as Garmin vivosmart 4 Tracker. This watch will be used to measure the deep sleep, REM sleep and wake-up time in hours.
To assess the efficacy of the Investigational Product (IP) from baseline on | Day 28
  The change in sleep index through the global scores of the Pittsburgh Sleep Quality Index (PSQI)
To assess the efficacy of the Investigational Product (IP) from baseline on | Day 21
  The change in sleep index through the global scores of the Pittsburgh Sleep Quality Index (PSQI)
To assess the efficacy of the Investigational Product (IP) from baseline on | Day 14
  The change in sleep index through the global scores of the Pittsburgh Sleep Quality Index (PSQI)
To assess the efficacy of the Investigational Product (IP) from baseline on | Day 7
  The change in sleep index through the global scores of the Pittsburgh Sleep Quality Index (PSQI)
To assess the efficacy of the Investigational Product (IP) from baseline on | Day 28
  Mood using POMS-A (Profile of Moods States - Abbreviated version)
To assess the efficacy of the Investigational Product (IP) from baseline on | Day 21
  Mood using POMS-A (Profile of Moods States - Abbreviated version)
To assess the efficacy of the Investigational Product (IP) from baseline on | Day 14
  Mood using POMS-A (Profile of Moods States - Abbreviated version)
To assess the efficacy of the Investigational Product (IP) from baseline on | Day 7
  Mood using POMS-A (Profile of Moods States - Abbreviated version)
To assess the efficacy of the Investigational Product (IP) from baseline on | Day 28
  Salivary cortisol levels immediately after waking up in the morning (before doing any activity)
To assess the efficacy of the Investigational Product (IP) from baseline on | Day 21
  Salivary cortisol levels immediately after waking up in the morning (before doing any activity)
To assess the efficacy of the Investigational Product (IP) from baseline on | Day 14
  Salivary cortisol levels immediately after waking up in the morning (before doing any activity)
To assess the efficacy of the Investigational Product (IP) from baseline on | Day 7
  Salivary cortisol levels immediately after waking up in the morning (before doing any activity)

CONTACTS AND LOCATIONS:
Locations (6):
- India (6):
  - V.S. General Hospital, Ahmedabad, Gujarat
  - Aman Hospital and Research Center, Vadodara, Gujarat
  - Poojan Multispeciality Hospital, Ahmedabad, Maharashtra
  - Shree Ashirwad Hospital, Dombivali, Maharashtra
  - Sai Cititcare, Ulhasnagar, Maharashtra
  - Maharaja Agrasen Superspeciality Hospital, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: Undecided